CLINICAL TRIAL: NCT04015596
Title: Double-Blind, Randomized, Placebo-Controlled Trial of Naproxen Sodium for the Treatment of Obsessive Compulsive Symptoms in Pediatric Autoimmune Neuropsychiatric Disorder Associated With Streptococcal Infections (PANDAS)
Brief Title: Trial of Naproxen Sodium for the Treatment of OCD in Children With PANDAS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Kyle A Williams, MD, PhD, Director, Pediatric Neuropsychiatry and Immunology Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019P000623
Record Dates: First submitted 2019-06-11; First posted 2019-07-11 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2023-03

CONDITIONS: PANDAS; Anxiety Disorder; Autoimmune Diseases; Obsessive-Compulsive Disorder
Keywords: PANDAS; Children; Obsessive-Compulsive Disorder; Anxiety; NSAID
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Anxiety Disorders; Autoimmune Diseases; Obsessive-Compulsive Disorder | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intervention (Experimental): Participants receive Naproxen Sodium.
  Interventions: Drug: Naproxen Sodium
- Placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Naproxen Sodium — Dosed by weight (10mg/kg), twice daily, for 8 weeks
  Arms: Intervention
Other: Placebo — Participants take placebo pills twice daily, for 8 weeks.
  Arms: Placebo

SUMMARY:
This project aims to rigorously evaluate a potential treatment for inflammation-related Obsessive-Compulsive Disorder (OCD) symptoms in children. To accomplish this goal, the investigators will conduct a double-blind, randomized, placebo-controlled trial of Naproxen Sodium, a nonsteroidal anti-inflammatory drug (NSAID) in participants diagnosed with Pediatric Autoimmune Neuropsychiatric Disorder Associated with Streptococcal infections (PANDAS). This research fills a gap in the empirical evidence base for the treatment of PANDAS, and will add to a growing literature of empirically-derived practices for PANDAS.

DETAILED DESCRIPTION:
The investigators propose to systematically evaluate the effects of naproxen sodium on anti-obsessional and behavioral improvement and conduct the first randomized controlled trial of naproxen sodium in the treatment of children with PANDAS. The study will involve an 8-week, double-blinded randomized controlled trial to evaluate the efficacy of naproxen sodium (10mg/kg, by mouth, twice a day) versus placebo to treat OCD symptoms in children with PANDAS. The investigators will acquire completed data on 44 children with PANDAS for this pilot study (i.e., 22 randomized to active treatment; 22 randomized to placebo). Outcome will be assessed comparing pre- and post-treatment OCD symptom severity using a standardized, clinician-administered interview assessing OCD symptoms by an independent rater blind to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. significantly interfering Obsessive-Compulsive Disorder (OCD) symptoms
2. ages 6- to 15-years-old
3. new-onset of OCD symptoms within the previous 18 months
4. sufficient fluency of English to understand study staff, procedures and questionnaires,
5. able to take medication in pill form
6. parent/legal guardian who can provide informed consent.

Patients must also meet all criteria for PANDAS, which are:

1. prepubertal symptom onset
2. acute onset of symptoms (from no/minimal symptoms to maximum severity within 24-48 hours) and/or an episodic (relapsing-remitting) course
3. temporal association between symptomatic periods and infections with Group A Streptococcus (GAS) infection
4. presence of neurological abnormalities (e.g. handwriting deterioration, choreiform movements).

The onset/exacerbation of OCD symptoms must also be accompanied by at least three of the following clinical signs and symptoms, including:

1. Markedly increased level of anxiety, particularly new onset of separation anxiety
2. Emotional lability, irritability, aggressive behavior and/or personality change
3. Sudden difficulties with concentration or learning
4. Developmental regression ("baby-talk", temper tantrums).
5. Sleep disorder (insomnia, night terrors, refusal to sleep alone)
6. Handwriting deterioration or other sign of motoric dysfunction (including new onset of motor hyperactivity, presence of choreiform finger movements, pronator drift or truncal instability)
7. Urinary frequency or increased urge to urinate; daytime or night-time secondary enuresis

These co-occurring symptoms must be "severe" or "dramatic" and proceed from no/minimal symptoms to maximum severity within the same 24-48 hour interval during which the OCD symptoms arose. In addition to these inclusion criteria, PANDAS subjects will be required to provide documentation of a positive GAS infection via medical records. As the time between a documented GAS infection and the onset of PANDAS symptoms has not been defined in the PANDAS diagnostic criteria, the investigators will use a guideline of approximately six weeks or less between a documented GAS infection and the onset of OCD symptoms for inclusion into the study.

Exclusion Criteria:

1. child who is acutely psychotic or suicidal
2. child has a serious neurological disorder or impairment (e.g. brain damage, blindness, deafness), an intellectual disability, or autism
3. history of immune modulating therapies for OCD/PANDAS symptoms
4. pre-existing liver, kidney, GI bleeding or clotting disorders (GFR <75 mL/min/1.73m2)
5. history of ulcers in the digestive system
6. history of restricted fluid intake, as this could exacerbate side effects
7. concurrent antibiotic treatment or antibiotic treatment within one-week of baseline
8. pregnant or becomes pregnant
9. currently engaged in an intensive outpatient cognitive behavioral treatment program (more than weekly)
10. concurrent selective serotonin reuptake inhibitor (SSRI) or other psychoactive medication treatment except and unless the dose has been stable for at least 6 weeks (i.e. no recent titration, initiation, or change in dosage)
11. concurrent medications that do not meet the above criteria (e.g., other psychotropic medications or anti-inflammatory agents)
12. history of severe asthma or currently uncontrolled asthma

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Children's Yale-Brown Obsessive-Compulsive Scale, 2nd Edition (CY-BOCS-II) | Pre- to Post-8 week treatment
  The CY-BOCS-II is a clinician-rated measure to assess obsessive-compulsive symptom severity. This results in two subscale total scores, Obsessions and Compulsion, each ranging from 0-25, with a higher score indicating more symptom severity. These subscale scores are summed to provide a total score, ranging from 0 to 50, that is used to measure overall OCD symptom severity.
Children's Yale-Brown Obsessive-Compulsive Scale, 1st Edition (CY-BOCS-I) | Pre- to Post-8 week treatment
  The CY-BOCS-I is a clinician-rated measure to assess obsessive-compulsive symptom severity. This results in two subscale total scores, Obsessions and Compulsion, each ranging from 0-20, with a higher score indicating more symptom severity. These subscale scores are summed to provide a total score, ranging from 0 to 40, that is used to measure overall OCD symptom severity.

SECONDARY OUTCOMES:
Changes in C reactive protein pre- and post-treatment between groups | Pre- to Post-8 week treatment
  C reactive protein (CRP, mg/L) will be obtained from pre- and post-blood draws and will be compared between groups.
Changes in erythrocyte sedimentation rate pre- and post-treatment between groups | Pre- to Post-8 week treatment
  Erythrocyte sedimentation rate (ESR, mm/h) will be obtained from pre- and post-blood draws and will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No